CLINICAL TRIAL: NCT05474976
Title: Compliance With Gluten-Free Diet and Affecting Factors in Adolescents With Celiac Disease During the Covid-19 Pandemic
Brief Title: Compliance With Gluten-Free Diet and Affecting Factors in Adolescents With Celiac Disease
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Ayla Irem Aydin, Principal Investigator, PhD, RN, Uludag University
Other Study IDs: 517517518
Record Dates: First submitted 2022-07-20; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Celiac Disease in Adolescents; Gluten-Free Diet in the Covid-19 Process
Keywords: Adolescence; Celiac Disease; gluten free diet
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Celiac is a chronic autoimmune disease that is treated with a gluten-free diet. Adolescents with celiac disease were affected differently by the restrictions during the COVID-19 pandemic. The aim of this study was to determine the compliance with a gluten-free diet during in adolescents with celiac disease during the Covid-19 pandemic and identify the associated factors.

The sample of this study consisted of 85 adolescents in the 10-19 age group diagnosed with celiac disease. Research data were collected by online questionnaires (Google Forms) between January and April 2022. Sociodemographic and disease-related data of adolescents who were compliant and those who were non-compliant with a gluten-free diet during the COVID-19 pandemic were compared.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 10-19 age group,
* Being diagnosed with celiac disease according to the revised ESPGHAN criteria,
* Following a gluten-free diet for at least 6 months before the COVID-19 lockdown,
* Consenting to participate in the study by the adolescents and their parents.

Exclusion Criteria:

-Having any cognitive or mental disorders.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population of this cross-sectional study of adolescents diagnosed with celiac disease in the 10-19 age group, registered to an association. Study sample of 85 participants who met the inclusion criteria and agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Adolescents with celiac disease adherence to their diet | 4 month
  In this study, dietary compliance of adolescents with celiac disease was examined using the Gluten-Free Diet Compliance Form.

SECONDARY OUTCOMES:
The effects of the pandemic on the gluten-free diet | 4 month
  The Factors Affecting Gluten-Free Diet Compliance form was used to determine the factors affecting adolescents' adherence to a gluten-free diet during the Covid-19 pandemic period.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla İrem Aydın, Phd, Principal Investigator — Uludag University
Locations (1):
- Bursa Uludağ University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It can be shared if there is a request for sharing.